CLINICAL TRIAL: NCT04739982
Title: A Lead-in Study Evaluating Mobile Game Based Therapy Among Children With Autism
Brief Title: A Lead-in Study Evaluating Efficacy of GuessWhat Mobile App Therapy for Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Principal Investigator, Dennis Paul Wall, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 60181; 5R01LM013364-03 (NIH)
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: digital health; mhealth; autism; intervention; behavioral therapy
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment (Experimental): The GuessWhat app is a charades style game and app that engages parent and child in fluid social interaction where the parent must guess what the child is acting out based on the prompt shown on the phone screen. Participants will use their own personal phone to download the study app. Parent and child will be encouraged to play using the emojis and emotion game mode at least 3 individual game sessions per week. Parents are asked to play GuessWhat with their child 3-4 times per week for 4 weeks.
  Interventions: Device: GuessWhat Mobile App
- Treatment as Usual (No Intervention): Participants in control group will continue their treatment as usual.

INTERVENTIONS:
Device: GuessWhat Mobile App — The GuessWhat app is a charades style game and app that engages parent and child in fluid social interaction where the parent must guess what the child is acting out based on the prompt shown on the phone screen. Participants will use their own personal phone to download the study app. Parent and child will be encouraged to play using the emojis and emotion game mode at least 3 individual game sessions per week. Parents are asked to play GuessWhat with their child 3-4 times per week for 4 weeks.
  Arms: Treatment

SUMMARY:
The following study aims to assess the efficacy, safety data, and best outcome measurements of the mobile game platform, GuessWhat, in delivering behavioral therapy to children with Autism Spectrum Disorder (ASD). GuessWhat is a mobile application (available for free for iOS and Android) which contains a suite of games: pro-social charades, emotion guessing, and quiz. Participant families will use their personal smartphones to download the app and play it with their child according to a predetermined regimen.

DETAILED DESCRIPTION:
The following study aims to understand the efficacy and safety of the mobile game platform, GuessWhat, in delivering behavioral therapy to children with Autism Spectrum Disorder (ASD). GuessWhat is a mobile application (available for free for iOS and Android) which contains a suite of games: pro-social charades, emotion guessing, and quiz. Participant families will use their personal smartphones to download the app and play it with their child according to a predetermined regimen. The study will enroll parents who are at least 18 years old and have a child between 3 and 12 years old with a formal ASD diagnosis. Parents will be asked to complete two clinical outcome measure questionnaires immediately prior to and up to 1 week after playing GuessWhat with their child 3 times per week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Parent who is at least 18 years old of child with autism.
2. Child with autism is between 3 and 12 years old at time of baseline data collection.

Exclusion Criteria:

1. Parent is unable to read English.
2. Parent does not have an Android or iOS smartphone compatible with GuessWhat App--the app will be available on Android after further development and we will notify interested families when it becomes available.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 541 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis P Wall, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: within 1 year after study completion

REFERENCES:
- See also: study sign up page — https://redcap.link/AutismSmartphoneStudy
- See also: GuessWhat Website — https://guesswhat.stanford.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between June 1, 2021 and July 1, 2022 using emails and online research listings.
Period: Overall Study
Arm/Group | Treatment | Treatment as Usual
Started | 322 | 219
Completed Week 4 Survey | 127 | 149
Completed | 127 | 149
Not Completed | 195 | 70
Not completed — Lost to Follow-up | 176 | 65
Not completed — Withdrawal by Subject | 19 | 0
Not completed — Protocol Violation | 0 | 5

BASELINE CHARACTERISTICS:
Population: Participants who completed follow-up survey at week 4
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Treatment as Usual | Total
Number analyzed (Participants) | 127 | 149 | 276
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 127 | 149 | 276
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 7.89 [3 to 12] | 7.47 [3 to 12] | 7.66 [3 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 64
  Male | 94 | 118 | 212
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Some participants may be counted twice as we allowed for multi-select in out form for race/ethnicity.
  Participants
    American Indian or Alaska Native | 1 | 6 | 7
    Black or African American | 19 | 18 | 37
    East Asian | 7 | 13 | 20
    Hispanic or Latino | 18 | 23 | 41
    Middle Eastern | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
    South Asian | 5 | 15 | 20
    Unknown / Not Listed | 34 | 42 | 76
    Caucasian/White | 47 | 47 | 94
Vineland Adaptive Behavior Scales-3 Socialization Subscale Standard Score [Mean (Standard Deviation); unit: score on a scale] — Vineland Adaptive Behavior Scales, 3rd edition (VABS-3) Socialization subscale of the Parent/Caregiver Comprehensive form will be administered online to the parents. Scores from the socialization domain of the VABS-III reflects one's functioning in social situations. The socialization subscale is up to 112 items depending on age and development, where raw scores are converted to IQ-type standard scores with mean 100 and standard deviation of 15, and factor in age equivalents, growth scale values, and higher scores indicate better adaptive functioning. The range for each subscale is 20 to 140.
  score on a scale | 72.30 (16.68) | 66.97 (18.42) | 69.42 (17.84)
Parental Stress Scale Score [Mean (Standard Deviation); unit: score on a scale] — The Parental Stress Scale is an 18-item parent report scale that evaluates the extent of parent stress. Scores range from 18-90, where higher scores indicate a higher level of Parental stress.
  score on a scale | 47.06 (9.13) | 47.95 (9.81) | 47.54 (9.40)
Mobile Autism Risk Assessment [Mean (Full Range); unit: score on a scale] — The Mobile Autism Risk Assessment (MARA) is an electronically administered, 7-question autism spectrum disorder (ASD) screening tool to triage those at highest risk for ASD. Scores range from -10 to 10, with negative scores indicating high risk, and positive scores suggesting low risk for ASD.
  score on a scale | -3.39 [-9.28 to 6.434] | -3.82 [-9.28 to 5.684] | -3.62 [-9.28 to 6.434]

OUTCOME MEASURES:

1. Primary Outcome: Change in Parent Reported Socialization Based on the Vineland Adaptive Behavior Scales 3rd Edition (VABS-3) Parent/Caregiver Socialization Subscale, From Baseline to Week 4
Description: Vineland Adaptive Behavior Scales, 3rd edition (VABS-3) Socialization subscale of the Parent/Caregiver Comprehensive form will be administered online to the parents. Scores from the socialization domain of the VABS-III reflects one's functioning in social situations. The socialization subscale is up to 112 items depending on age and development, where raw scores are converted to IQ-type standard scores with mean 100 and standard deviation of 15, and factor in age equivalents, growth scale values, and higher scores indicate better adaptive functioning. The range for each subscale is 20 to 140.
Time Frame: Baseline (Week 0), Week 4
Population: Participants who completed follow-up survey at week 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Treatment | Treatment as Usual
Number analyzed (Participants) | 127 | 149
score on a scale | .56 (.98) | .23 (.96)
Statistical Analysis 1: Comparison: Treatment vs Treatment as Usual; Test type: Superiority; p = .41, t-test, 1 sided — An independent samples t-test was conducted to compare the change in baseline and follow-up scores of treatment and treatment as usual participants; Degrees of freedom=274 Significance level=.05; Cohen's D = .03, 95% CI 2-sided [-.21 to .27], Standard Error of Mean 1.36

2. Secondary Outcome: Change in Parental Stress Scale - From Baseline to Week 4
Description: The Parental Stress Scale is an 18-item parent report scale that evaluates the extent of parent stress. Scores range from 18-90, where higher scores indicate a higher level of Parental stress. Parents completed this survey, but were not considered to be enrolled in the study.
Time Frame: Baseline (Week 0), Week 4
Population: Participants who completed follow-up survey at week 4
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment | Treatment as Usual
Number analyzed (Participants) | 127 | 149
units on a scale | -5.18 (.76) | -7.01 (1.17)
Statistical Analysis 1: Comparison: Treatment vs Treatment as Usual; Test type: Superiority; p = .095, t-test, 1 sided; Cohen's D = .153, 95% CI 2-sided [-.08 to .39], Standard Error of Mean 1.45

3. Secondary Outcome: GuessWhat App Usage Data
Description: App usage data by participants (children) comprised of number of MojiMatch and Charades Games started.
Time Frame: Baseline through week 4 (assessed at week 4)
Population: Participants with available data. Only the Treatment Group is included in the analysis, as the Treatment as Usual Group did not use the app.
Measure: Mean (Standard Deviation); unit: number of games
Arm/Group | Treatment
Number analyzed (Participants) | 90
number of games | 15.77 (25.43)

4. Secondary Outcome: Change in Emotion Recognition From Baseline to Week 4
Description: Study team used an image based emotion recognition task where participants (children) will select the emotion that corresponds to an emotional facial image in the form of a GIF (Graphics Interchange Format) image. Participants select 1 of 8 available Ekman emotion labels for 16 facial emotional image stimuli presented in random order. Correct responses will be measured against a predetermined majority rules consensus of the emotional content of the GIFs. Scores range from 0 (no emotional image stimuli correctly identified) to 16 (all correctly identified).
Time Frame: Baseline (Week 0), Week 4
Population: Participants with available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Treatment as Usual
Number analyzed (Participants) | 97 | 102
score on a scale | -.37 (4.34) | -1.12 (3.42)
Statistical Analysis 1: Comparison: Treatment vs Treatment as Usual; Test type: Superiority; p = .09, t-test, 1 sided; Cohen's D = .19, 95% CI 2-sided [-.09 to .47], Standard Error of Mean .55

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Treatment | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/322 | 0/219
Serious Adverse Events (participants affected / at risk) | 0/322 | 0/219
Other Adverse Events (participants affected / at risk) | 0/322 | 0/219

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT04739982/Prot_SAP_002.pdf
  • Informed Consent Form (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT04739982/ICF_001.pdf